CLINICAL TRIAL: NCT05142618
Title: Pilot Trial of Abdominal Core Rehabilitation To Improve Outcomes After Ventral Hernia Repair
Acronym: ABVENTURE-P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ajit Chaudhari, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021H0336; R01DK131207 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-12-02 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Ventral Hernia; Hernia; Herniorrhaphy; Abdominal Wall; Postoperative Period; Physical Therapy Modalities
Keywords: ventral hernia repair; abdominal core health; physical therapy
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Post-operative Instructions (Active Comparator): Participants in the control group will be told upon post-operative discharge that they should follow the post-operative instructions.
  Interventions: Other: Post-operative Precautions
- Supervised Physical Therapy (Experimental): Participants in the physical therapy group will be scheduled for visits to the physical therapy clinic beginning two weeks after surgery, and will undergo supervised physical therapy treatments approximately twice per week for eight weeks according to a standardized evidence-based post-operative abdominal core surgery rehabilitation program.
  Interventions: Other: Supervised Physical Therapy

INTERVENTIONS:
Other: Supervised Physical Therapy — The twice-per-week 8-week course of supervised physical therapy begins 2 weeks after surgery. It targets abdominal core function through progressive muscle retraining and strengthening, and patient-specific posture and body mechanics education.
  Arms: Supervised Physical Therapy
Other: Post-operative Precautions — This intervention includes standard of care post-operative instructions typically given to patients undergoing ventral hernia repair across the world. These include limiting strenuous physical activity and a lifting restriction of no more than 10 pounds for 6 weeks. Binder use is also encouraged for 4-6 weeks after the operation.
  Arms: Standard Post-operative Instructions

SUMMARY:
This study aims to evaluate the potential role of physical therapy in improving outcomes after ventral hernia repair.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will perform assessments of several activities of daily living and complete several surveys detailing their pre-surgical abilities, quality of life, and pain. Immediately after their surgical procedure, patients will be randomized in a single-blind manner (investigator) in a 1:1 ratio to supervised physical therapy (8 weeks, twice weekly) or standard post-surgical precautions. Assessments and surveys will be repeated by the blinded investigator at 30 days, 10 weeks, 6 months, and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria

* Ages 18+
* Diagnosis of ventral hernia
* Scheduled for elective ventral hernia repair
* Independent functional status
* Transverse hernia width of 2cm or greater

Exclusion Criteria

* Previously diagnosed movement or balance disorder
* Use of ambulatory assistive device (walker or cane)
* Not currently undergoing or planning to undergo physical therapy or other skilled exercise intervention supervised by a medical rehabilitation professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Five times sit-to-stand time | Baseline before surgery, 10 weeks after surgery
  From a standard chair, stand and sit back down five times in immediate succession as quickly as possible.
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function | Baseline before surgery, 10 weeks after surgery
  Computer-adaptive patient-reported questionnaire asking questions about physical function.
Change from Baseline in Quiet unstable sitting test | Baseline before surgery, 10 weeks after surgery
  Sit on an inflated cushion that creates an unstable surface for 60 seconds with eyes closed and arms crossed while counting to a metronome.

SECONDARY OUTCOMES:
Change in Hernia related quality of life survey from baseline | baseline before surgery, 10 weeks after surgery
  Patient-reported questionnaire asking questions about abdominal wall function including activities of daily living, independent mobility, and mental health.
Change in Timed Up-And-Go time from baseline | baseline before surgery, 10 weeks after surgery
  Starting seated in a standard chair, stand, walk forward 3 m, turn 180 deg, walk back to chair, sit down. Do all of these as quickly as can be done safely.
Change from baseline in International Physical Activity Questionnaire - Short Form | baseline before surgery, 10 weeks after surgery
  Self-reported physical activity questions spanning sedentary behavior, job activity, transportation activity, household activity, and recreational activity.
Change from baseline in Tampa Scale of Kinesiophobia - Short Form | baseline before surgery, 10 weeks after surgery
  Self-reported questions on how fear affects desire and ability to perform physical activities.
Hernia recurrence inventory | 1 year after surgery
  Patient-reported questionnaire asking questions regarding a recurrence of the hernia based on pain and presence of a physical bulge.
Change in Hernia related quality of life survey from baseline | baseline before surgery, 1 year after surgery
  Patient-reported questionnaire asking questions about abdominal wall function including activities of daily living, independent mobility, and mental health.
Change in Timed Up-And-Go time from baseline | baseline before surgery, 1 year after surgery
  Starting seated in a standard chair, stand, walk forward 3 m, turn 180 deg, walk back to chair, sit down. Do all of these as quickly as can be done safely.
Change from baseline in International Physical Activity Questionnaire - Long Form | baseline before surgery, 1 year after surgery
  Self-reported physical activity questions spanning sedentary behavior, job activity, transportation activity, household activity, and recreational activity.
Change from baseline in Tampa Scale of Kinesiophobia - Short Form | baseline before surgery, 1 year after surgery
  Self-reported questions on how fear affects desire and ability to perform physical activities.
Change from Baseline in Five times sit-to-stand time | baseline before surgery, 1 year after surgery
  From a standard chair, stand and sit back down five times in immediate succession as quickly as possible.
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function | baseline before surgery, 1 year after surgery
  Computer-adaptive patient-reported questionnaire asking questions about physical function.
Change from Baseline in Quiet unstable sitting test | baseline before surgery, 1 year after surgery
  Sit on an inflated cushion that creates an unstable surface for 60 seconds with eyes closed and arms crossed while counting to a metronome.

OTHER OUTCOMES:
Change in Hernia related quality of life survey from baseline | baseline before surgery, 30 days after surgery
  Patient-reported questionnaire asking questions about abdominal wall function including activities of daily living, independent mobility, and mental health.
Change in Timed Up-And-Go time from baseline | baseline before surgery, 30 days after surgery
  Starting seated in a standard chair, stand, walk forward 3 m, turn 180 deg, walk back to chair, sit down. Do all of these as quickly as can be done safely.
Change from baseline in International Physical Activity Questionnaire - Short Form | baseline before surgery, 30 days after surgery
  Self-reported physical activity questions spanning sedentary behavior, job activity, transportation activity, household activity, and recreational activity.
Change from baseline in Tampa Scale of Kinesiophobia - Short Form | baseline before surgery, 30 days after surgery
  Self-reported questions on how fear affects desire and ability to perform physical activities.
Change from Baseline in Five times sit-to-stand time | baseline before surgery, 30 days after surgery
  From a standard chair, stand and sit back down five times in immediate succession as quickly as possible.
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function | baseline before surgery, 30 days after surgery
  Computer-adaptive patient-reported questionnaire asking questions about physical function.
Change from Baseline in Quiet unstable sitting test | baseline before surgery, 30 days after surgery
  Sit on an inflated cushion that creates an unstable surface for 60 seconds with eyes closed and arms crossed while counting to a metronome.
Change in Hernia related quality of life survey from baseline | baseline before surgery, 6 months after surgery
  Patient-reported questionnaire asking questions about abdominal wall function including activities of daily living, independent mobility, and mental health.
Change in Timed Up-And-Go time from baseline | baseline before surgery, 6 months after surgery
  Starting seated in a standard chair, stand, walk forward 3 m, turn 180 deg, walk back to chair, sit down. Do all of these as quickly as can be done safely.
Change from baseline in International Physical Activity Questionnaire - Long Form | baseline before surgery, 6 months after surgery
  Self-reported physical activity questions spanning sedentary behavior, job activity, transportation activity, household activity, and recreational activity.
Change from baseline in Tampa Scale of Kinesiophobia - Short Form | baseline before surgery, 6 months after surgery
  Self-reported questions on how fear affects desire and ability to perform physical activities.
Change from Baseline in Five times sit-to-stand time | baseline before surgery, 6 months after surgery
  From a standard chair, stand and sit back down five times in immediate succession as quickly as possible.
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) - Physical Function | baseline before surgery, 6 months after surgery
  Computer-adaptive patient-reported questionnaire asking questions about physical function.
Change from Baseline in Quiet unstable sitting test | baseline before surgery, 6 months after surgery
  Sit on an inflated cushion that creates an unstable surface for 60 seconds with eyes closed and arms crossed while counting to a metronome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared with other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05142618/ICF_000.pdf